CLINICAL TRIAL: NCT07054385
Title: I-CARE-Rural Pilot: Remote Digital Intervention for Rural-Dwelling Dementia Caregivers
Brief Title: I-CARE Rural Pilot: Intervention for Rural-Dwelling Dementia Caregivers
Acronym: I-CARE-Rural-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Holden (Other)
Responsible Party: Sponsor-Investigator, Richard Holden, Principal Investigator, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 27397
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-06

CONDITIONS: Caregiver Burden; Alzheimer Disease
Keywords: Alzheimer disease and related dementias; Caregiver; Caregiver Burden; Behavioral and psychological symptoms of dementia; Rural
MeSH Terms: conditions — Caregiver Burden; Alzheimer Disease; Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive the Brain CareNotes app or an attention control app.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, primary investigator and outcome assessor will be masked to the app assignment (Brain CareNotes vs Attention Control App). The participant will be aware of the treatment received but is masked to whether the app they are assigned is the intervention versus control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain CareNotes App (Experimental): The Brain CareNotes mobile telehealth app is used by unpaid caregivers for BPSD management. It includes remote communication with an external human support person-a care coach-as well as features for users to independently perform health-related activities.
  Interventions: Behavioral: Brain CareNotes
- Attention Control App (Active Comparator): Dementia Guide Expert provides education only and no interactive BPSD management support, coaching, assessment, or external response. It contains "evidence-based expert information on what dementia is, types, contributing factors, risks, symptoms, stages, diagnosis, tests, treatment, management, communication techniques, and links to resources and support services."
  Interventions: Behavioral: Dementia Guide Expert

INTERVENTIONS:
Behavioral: Brain CareNotes — The Brain CareNotes mobile telehealth app is used by unpaid caregivers for BPSD management. It includes remote communication with an external human support person-a care coach-as well as features for users to independently perform health-related activities.
  Arms: Brain CareNotes App
Behavioral: Dementia Guide Expert — Dementia Guide Expert provides education only and no interactive BPSD management support, coaching, assessment, or external response. It contains "evidence-based expert information on what dementia is, types, contributing factors, risks, symptoms, stages, diagnosis, tests, treatment, management, communication techniques, and links to resources and support services."
  Arms: Attention Control App

SUMMARY:
The purpose of this study is to assess feasibility and to estimate efficacy of our app "Brain CareNotes" for dementia caregivers who reside in a rural setting (as defined by RUCA codes 4 through 10). The Brain CareNotes app is designed to reduce informal caregiver burden of those caring for individuals with Alzheimer's disease and related dementias (ADRD) and behavioral and psychological symptoms of dementia (BPSD) of individuals with ADRD. The study will enroll up to 60 rural caregivers of community-dwelling individuals living with ADRD. Caregivers will be randomized to use the Brain CareNotes app or an attention control education-only app for six months, with usage reminders.

DETAILED DESCRIPTION:
This study will evaluate the feasibility and estimate the effect of Brain CareNotes on caregiver burden and patient BPSD. The study will enroll up to 60 rural-dwelling caregivers. Participants will be randomized to use the Brain CareNotes app or an attention control education-only app (Dementia Guide Expert) for six months.

The primary objective is to evaluate the feasibility of Brain CareNotes, as assessed by caregiver-reported a) usability, as assessed by the 10-item Simplified System Usability Scale and b) acceptance as assessed by the 4-item Behavioral Intention questionnaire.

The secondary objective is to estimate the effect of Brain CareNotes on a) caregiver burden and b) patient BPSD at six months, compared to attention control. These outcomes are calculated using the caregiver-reported Neuropsychiatric Inventory (NPI): the NPI caregiver distress sub-score measures caregiver burden and the NPI total score measures patient BPSD. The investigators will obtain NPI responses from caregivers at baseline, three, and six months.

Exploratory objectives are to estimate the effect of Brain CareNotes on a) caregiver depressive symptoms and b) patient and caregiver acute care utilization at six months; and to examine early effects at three months on c) the usability and acceptance of Brain CareNotes, and d) caregiver burden and BPSD. Caregiver depressive symptoms will be assessed by the Patient Health Questionnaire-9 (PHQ-9), administered at baseline, three, and six months. Acute care utilization data will be obtained from self-reports to identify both caregivers' and patients' hospital and emergency visits that occurred within six months of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified primary unpaid rural (RUCA Code of 4-10) caregiver of a person diagnosed with ADRD (at any stage) who are:
* Receiving primary care and
* Community-dwelling;
* English literate;
* Age ≥ 18 years

Exclusion Criteria:

* Care recipient is a permanent resident of an extended care facility (nursing home);
* Involvement in another clinical trial that would prevent or interfere with study objectives;
* Sensory or other impairment prohibiting the use of a mobile touchscreen device or other study activity (after correction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
App Usability | Six Months
  10-item standardized survey of user-reported technology usability, based on revised System Usability Scale, with scale score computed ranging from 0-100, with 100 indicating highest possible perceived usability.
App Acceptability | Six Months
  A 4-item questionnaire assessing a user's intention to use a technology in the near future. Scores range from 0-24 with a high score representing greater intention to use the technology.

SECONDARY OUTCOMES:
Patient BPSD | Six Months
  Behavioral (e.g. agitation, aggression, wandering) and psychological (e.g. delusions, hallucinations) symptoms of dementia as measured by the Neuropsychiatric Inventory (NPI). The NPI is a 12-item questionnaire. The total score is calculated by adding the product of the frequency and severity of those 12 items. A score of 0 would indicate that no symptoms are present while a score of 144 would indicate that all symptoms are present at the highest level of frequency and severity.
Caregiver Burden | Six Months
  The burden experienced by caregivers caused by their caregiving responsibilities measured by the Neuropsychiatric Inventory (NPI) caregiver distress sub-score. The distress score is calculated by adding the distress score for each of the 12 items of the NPI. A score of 0 would indicate that the BPSD cause no distress while a score of 60 would indicate that each symptom causes severe distress for the caregiver.

OTHER OUTCOMES:
Caregiver Depressive Symptoms | Six Months
  Caregiver depression as measured by the Patient Health Questionnaire (PHQ)-9. The PHQ-9 is a 9-item questionnaire using a 0-3 rating scale. Scores range from 0-27. A total score of 0 represents no depression, while score of 5, 10, 15, and 20 serve as cut points for mild, moderate, moderately severe, and severe depression, respectively.
Patient Acute Care Utilization | Six Months
  Patient visits to emergency rooms, hospitals, or inpatient diagnoses. Obtained from caregiver self-reports.
Caregiver Acute Care Utilization | Six Months
  Caregiver visits to emergency rooms, hospitals, or inpatient diagnoses. Obtained from caregiver self-reports.
Caregiver Self-Efficacy | Six Months
  Caregiver perceived self-efficacy as measured using the Revised Scale for Caregiving Self-Efficacy. It consists of 3 sections each with five items. Participants rank self-efficacy on a scale of 0-100 for each item, with a higher score representing greater confidence. Thus, a high total score represents greater self-efficacy.
Caregiver Social Support | Six Months
  Caregiver perceived social support measured using the Multidimensional Scale of Perceived Social Support (MSPSS). The MSPSS is a 12-item questionnaire using a 7-point Likert scale where 1 is very strongly disagree and 7 is very strongly agree. Scores range from 12-84. A low score represents minimal social support while a high score represents a great level of perceived social support.
App Use | Six Months
  Usage logs of app use over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan R Hill, PhD, Principal Investigator — Indiana University, Bloomington; Richard J Holden, PhD, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University Bloomington, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No